CLINICAL TRIAL: NCT03799393
Title: Buckle Me Up!: A Computerized, Individually-Tailored Emergency Department Discharge Intervention for Child Car Restraint Safety Education
Brief Title: Buckle Me Up!: A Digital Emergency Department Discharge Intervention for Child Car Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lifespan (Other)
Responsible Party: Principal Investigator, Almaz Dessie, Principal Investigator, Lifespan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2012-17
Record Dates: First submitted 2018-12-24; First posted 2019-01-10 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Safety Issues; Injuries; Car Accident
Keywords: injury prevention; car safety; car seats; booster seats; car restraints
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): The control group will receive a brief tablet-based questionnaire followed by standard, paper discharge instructions on car safety. Children ≥13 years old and above will answer questions themselves. They will complete a questionnaire on the usefulness of their discharge education.
  One week after discharge, participants will receive an automatic text message and/or email message with a link to a web-based survey that will assess: knowledge of appropriate car restraints and whether the parent/patient engaged in any behavioral changes regarding child car restraint.
  Interventions: Behavioral: Standard Printed Discharge Instructions
- Experimental/CIAS Group (Experimental): The Experimental/CIAS Group will receive a brief tablet-based questionnaire followed by the intervention - CIAS, an interactive tablet computer program that gives educational information customized to the patient's age and size. Children ≥13 years old will answer questions and interact with the program themselves. They will complete a questionnaire on the usefulness of their discharge education.
  One week after discharge, participants will receive an automatic text message and/or email message with a link to a web-based survey that will assess: knowledge of appropriate car restraints and whether the parent/patient engaged in any behavioral changes regarding child car restraint.
  Interventions: Behavioral: CIAS (Computer Intervention Authoring Software)

INTERVENTIONS:
Behavioral: CIAS (Computer Intervention Authoring Software) — This is a digital application that allows families to interact with a tablet computer to receive educational information customized to the patient's age and size. allows authors to develop screening, assessment, and intervention tools for patients without requiring new programming. The CIAS intervention is programmed using tailored branching logic to allow a custom path through the intervention based on the respondent's answers. Delivery of the intervention uses a two-dimensional avatar narrator character that mimics the conversational structure of person-delivered brief interventions.
  Arms: Experimental/CIAS Group
Behavioral: Standard Printed Discharge Instructions — Patients/families will receive standard, printed discharge instructions. This is a 5 page general document from our Injury Prevention Center that describes appropriate car restraint safety for all age groups, not specific to the child enrolled.
  Arms: Control Group

SUMMARY:
This study explores the utility of a tablet computer-based, individually-tailored application called Computer Intervention Authoring Software (CIAS) in the Emergency Department for discharge education on proper child car restraint safety. The investigators hypothesize that tablet-based, individually-tailored discharge instructions are more effective than current standard, one-size-fits-all, printed discharge instructions. This is a randomized, controlled, non-blinded trial of of children age 0-21 years old in the Emergency Department. Patients will be randomized to receive either (a) a brief tablet-based questionnaire followed by standard, paper discharge instructions or (b) a brief tablet-based questionnaire followed by the intervention - CIAS, a tablet-based computer program. One week after discharge, participants in both groups will receive an automatic text message and/or email message with a link to a web-based survey that will assess: knowledge of appropriate car restraints and whether the parent/patient engaged in any behavioral changes regarding child car restraint. These variables will be compared between the control and intervention groups.

DETAILED DESCRIPTION:
This study explores the utility of a tablet computer-based, individually-tailored technology called Computer Intervention Authoring Software (CIAS) in the Emergency Department for discharge education on proper child car restraint safety. The investigators hypothesize that tablet-based, individually-tailored discharge instructions are more effective than current standard, one-size-fits-all, printed discharge instructions. This is a randomized, controlled, non-blinded trial of a convenience sample of 200 children age 0-21 years old who present to the Hasbro Children's Hospital Emergency Department by car and have access to a smartphone and/or email. Patients will be randomized to receive either (a) a brief tablet-based questionnaire followed by standard, paper discharge instructions or (b) a brief tablet-based questionnaire followed by the intervention - CIAS, a computer program that allows families to interact with a tablet computer to receive educational information customized to the patient. Children 13 years old and above will answer questions themselves instead of having their parent/guardian answer for them. Both group will be offered information for the Lifespan Injury Prevention Center's Kohl's Car Seat Program. Both groups will complete a questionnaire on the usefulness of their discharge education. One week after discharge, participants in both groups will receive an automatic text message and/or email message with a link to a web-based survey that will assess: knowledge of appropriate car restraints and whether the parent/patient engaged in any behavioral changes regarding child car restraint. These variables will be compared between the control and intervention groups.

ELIGIBILITY:
Inclusion Criteria:

- Children age 0-21 years presenting to the children's emergency department for any chief complaint whose parent/guardian owns or has access to a car that the child rides in (or for adolescents 16 years or older, have access to a car themselves).

Exclusion Criteria:

* No access to email or a smart phone
* Adolescents with significant developmental delay
* Adolescents who are critically injured
* No parent/guardian present at time of enrollment

Max Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 295 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Demonstration of age-appropriate car restraint knowledge | one week after enrollment
  Rate of correct response to a post-intervention follow-up survey question regarding age appropriate car restraint for child in control group vs. intervention group.
Change in car restraint knowledge | one week after enrollment
  Change in rate of correct response pre-intervention vs. post-intervention compared between control group vs. intervention

SECONDARY OUTCOMES:
Actions taken related to car restraints | one week after enrollment
  Rate of parental self-report of actions taken related to changing use of car restraints on post-intervention follow-up survey. This will be a binary variable (NO action taken vs. YES action taken).
Rate of difference types of actions taken related to car restraints | one week after enrollment
  Rates of each specific type of actions taken will also be compared between control and intervention groups (e.g. percentage of subjects who purchased a new car restraint device in each group, percentage of patients that had car seat installation checked at a fire department in each group, etc).
Satisfaction with discharge education - CIAS | during intervention/enrollment
  For intervention group only - parent/patient satisfaction with education given on discharge based on score on Technology Posttrial Impressions Questionnaire. We will examine 13 individual components scored on an ordinal scale 1 to 5 (poor, fair, good, very good, excellent). Mean total score will be calculated.
Parental confidence in type of car restraint | one week after enrollment
  Change in parental confidence that child is in the correct type of car restraint, comparing pre- and post-intervention response according to the 1 to 5 ordinal scale:
  How confident are you that your child is in the right type of car restraint?
  1- not at all confident 2- 3- 4- 5- very confident
Parental confidence in car restraint installation | one week after enrollment
  Change in parental confidence that car restraint is correctly installed, comparing pre- and post-intervention response according to the 1 to 5 ordinal scale:
  How confident are you that your car restraint is installed correctly?
  1- not at all confident 2- 3- 4- 5- very confident
Parental confidence in buckling the car restraint | one week after enrollment
  Change in parental confidence that the child is correctly buckled in the car restraint, comparing pre- and post-intervention response according to the 1 to 5 ordinal scale:
  How confident are you that your child is correctly buckled into the car restraint?
  1- not at all confident 2- 3- 4- 5- very confident

CONTACTS AND LOCATIONS:
Overall Officials: Susan Duffy, MD, MPH, Study Director — Associate Professor
Locations (1):
- Hasbro Children's Hospital Emergency Department, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang AY, Leviter J, Baird J, Charles-Chauvet D, Frackiewicz LM, Duffy S, Dessie A. Buckle me up! A randomised controlled trial using a tablet-based emergency department intervention for child car safety education. Inj Prev. 2024 Jul 19;30(4):334-340. doi: 10.1136/ip-2023-044998. PMID 38302281